CLINICAL TRIAL: NCT06201377
Title: Analysis of Early Healing After the Use of Two Types of Sutures in Periodontal Surgery. A Pilot Study.
Brief Title: Analysis of Early Healing of Sutures in Periodontal Surgery
Acronym: Sutures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ana María García de la Fuente (Other)
Responsible Party: Sponsor-Investigator, Ana María García de la Fuente, Professor, University of the Basque Country (UPV/EHU)
Organization: University of the Basque Country (UPV/EHU) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2023/01
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Post-Surgical Complication; Periodontal Inflammation; Surgical Site Infection
Keywords: Surgical site infection; Periodontal surgery; Post-surgical pain; Post-surgical inflammation; periodontitis
MeSH Terms: conditions — Surgical Wound Infection; Pain, Postoperative; Periodontitis | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: We will perform the experimental (periodontal surgery where the suture of the flap will be an absorbable suture with clorhexidine) control technique (periodontal surgery where the suture of the flap will be an absorbable suture without clorhexidine) according to the randomization sequence.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant: Initially, the subject will not know which suture he/she has received, full information regarding the suture used, as well as the results obtained in his/her case, will be given at the last visit of the study.
  Observer: (R.E. Another periodontist, external to the intervention, will be in charge of recording the clinical parameters.) Analyst: (X. M. The statistician does not know to which treatment each variable corresponds.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture with chlorhexidine (Experimental): At the end of the surgical procedure, the flap will be sutured with an absorbable suture coated with chlorhexidine diacetate (NOVOSYN CHLORHEXIDINE)
  Interventions: Other: Periodontal Access Surgery+ Suture with chlorhexidine
- Suture without chlorhexidine (Active Comparator): At the end of the surgical procedure, the flap will be sutured with an absorbable suture coated without chlorhexidine diacetate (NOVOSYN)
  Interventions: Other: Periodontal Access Surgery+ Suture without chlorhexidine

INTERVENTIONS:
Other: Periodontal Access Surgery+ Suture with chlorhexidine — Periodontal conventional surgery will be performed as treatment of periodontal diseases in patients who present active periodontal pockets. At the end of the surgery, the surgeon will suture the flap with the absorbable polyglactin 910 suture coated with chlorhexidine (Novosyn Chlorhexidine). Standardized post-surgical recommendations will be followed.
  Other Names: Novosyn Clorhexidine
  Arms: Suture with chlorhexidine
Other: Periodontal Access Surgery+ Suture without chlorhexidine — Periodontal conventional surgery will be performed as treatment of periodontal diseases in patients who present active periodontal pockets. At the end of the surgery, the surgeon will suture the flap with the absorbable polyglactin 910 suture (Novosyn). Standardized post-surgical recommendations will be followed.
  Other Names: Novosyn
  Arms: Suture without chlorhexidine

SUMMARY:
The main objective is to analyze post-surgical periodontal healing after conventional periodontal surgery where an absorbable suture coated with clorhexidine (Novosyn Clorhexidine) versus conventional sutures without chlorhexidine (Novosyn) will be used a pilot randomized clinical study has been designed.

Up to authors´ knowledge until now there are no studies to evaluate periodontal healing after periodontal surgery in combination with this kind of sutures.

DETAILED DESCRIPTION:
A total of 60 patients will be included, where the unit of study will be each stitch, among the patients attending the Dental Clinic Service of the University of the Basque Country (UPV/EHU) who require surgical periodontal treatment.

The patients will be randomly divided into two groups: the control group using a conventional suture (n=30), and the test group using a suture coated with chlorhexidine diacetate (n=30).

Suture in the control group: absorbable suture of polyglactin 910 coated with polyglactin 370 + calcium stearate without chlorhexidine (NOVOSYN) Suture in the test group: absorbable suture of polyglactin 910 coated with polyglactin 370 + calcium stearate and chlorhexidine diacetate (NOVOSYN CHLORHEXIDINE) The primary variable in this study is post-surgical healing in both groups, which will be assessed using the healing index.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years-old
* Patients who have completed the basic periodontal phase and require surgical periodontal treatment for periodontal disease control.
* Plaque index (O'Leary et al.,1972) ≤20%.
* Bleeding index (Ainamo & Bay,1975) ≤20%.

Exclusion Criteria:

* Patients with systemic conditions contraindicating surgery
* Patients with allergy to chlorhexidine and/or o-cymen-5-ol
* Patients allergic to non-steroidal anti-inflammatory drugs (NSAIDs)
* Pregnant or breastfeeding women
* Patients with periodontal defects requiring regenerative surgery or mucogingival surgery/periodontal plastic therapy
* Patients who have taken antibiotics in the last 3months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Periodontal healing index (PQI) (Landry et al., 1988) | at 7 days, 14 days, 1 month and 2 months after surgery
  This periodontal healing index was described by Landy et al. in 1988. The index consists of the assessment of 5 clinical parameters (tissue color, bleeding on palpation, presence of granulation tissue, presence of suppuration, and healing of the surgical margin). The index will be from 1 to 5, where point 1 was defined as "healing way scarce" and point 5 such as "excellent healing" (Landry RG, Turnbull RS, Howley T. Effectiveness of benzydamine HCL in the treatment of periodontal post-surgical patients. Res Clin Forums. 1988; 10:105-118)

SECONDARY OUTCOMES:
Pre-surgical pain | The day of the surgical intervention
  This variable will be collected by means of a questionnaire included in the pain diary (called "UPV/EHU pain diary" Fernández Jiménez et al., 2021).The examiner will record whether the subject has had any regional head and neck pain in the last month prior to the operation and whether any pain was present in the immediate pre-surgical period (last 24 hours). If so, its intensity will be recorded (visual analogue scale (from 0 to 10, where 0 represents no pain and 10 represents the maximum pain known to the subject.
Clinical level of central sensitization of the subject (Subclinical, Medium, Moderate, Severe and Extreme) | Prior to surgery
  Prior to surgery a Central Sensitization Questionnaire (CSC) will be used (Cuesta-Vargas et al., 2016), in which each subject is asked about the frequency with which they perceive 25 symptoms and will be given a score of 0-4.
  This will finally establish a clinical level in a range of 0-100 (Subclinical: 0-29 points; Medium: 30-39; Moderate: 40-49; Severe: 50-59; Extreme: 60-100).
Post-surgical pain | At 7 days after the surgery
  The subject will be given a pain diary (PD) based on the VAS (Fernández-Jiménez et al., 2021) with instructions for its completion.
  The subject will be instructed to record their perception of post-surgical pain at 2 and 4 hours, then every 8 hours for the first 3 days and finally daily at the end of the day for a week or until remission. Specifically, the subject will record three variables: the greatest intensity of the pain (0-100), its duration (minutes or hours) and whether any analgesic treatment has been necessary (No or Yes: Which one?). This information will be recorded until the pain has subsided
Achievement of primary closure after suturing (in the surgical act). | The day of the surgery
  At each sutured site, the distance between the edges of the incision will be measured with a periodontal probe, being 0 the primary closure and from there we measure the mm of separation.
Surgery location information (location of suture, surgery time, surgeon´s experience) | The day of the surgery
  Location of the suture, indicating the teeth between which it is located, as well as the quadrant where it has been performed.
  Surgery time: Minutes elapsed from the start of anesthesia to the knotting of the last stitch.
  Surgeon's experience: number of previous periodontal surgeries performed by the surgeon and length of experience measured in months
Post-surgical complications (PSCs) | The day of the removal of sutures
  The presence or not of any Post-surgical complications (PSCs) that may occur, as well as their description.
Presence of Visible plaque on the suture | The day of the removal of sutures
  Presence of Visible plaque on the suture (dichotomous: yes / no) on the day of stich removal, which will be assessed prior to their removal, noting the value in vestibular, palatal or lingual.
Suture looseness | The day of the removal of sutures
  It will be measured in mm with a calibrated periodontal probe, to the nearest 0.5 mm. Prior to cutting the suture, this will be grasped with stitch removal forceps, and the distance from the suture knot to the gingival tissue shall be measured.
Pain on suture removal | The day of the removal of sutures
  Pain on suture removal (dichotomous: yes/no) on suture removal, in which we will record whether or not the patient reports discomfort on suture removal.
Cytological-histological analysis | The day of the removal of sutures
  The suture of each patient will be analyzed by a) performing cytological smears (Papanicolaou stain) of the material deposited on the suture and b) histologically studying the knot (Included in 10% neutrally buffered formalin solution and later embedded in paraffin. Then, 8 μm thick sections were performed, which were stained with hematoxylin and eosin). Both analyses will be examined under an optical microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Ana María García-De-La-Fuente, phD, Study Director — University of the Basque Country (UPV/EHU); Aitziber Fernández-Jiménez, phD, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (1):
- Department fo Stomatology, Faculty of Medicine and Nursery, University of the Basque Country, Leioa, Biscay, Spain

IPD SHARING:
Plan to Share IPD: Yes
A code will identify the data collected for the study and only the researcher will be able to relate them. The personal data will be treated with absolute confidentiality in accordance with the Data Protection Law and will remain in the patient's clinical history. The coded data will be included in a UPV/EHU´s file with reference number (ENFERMEDADES PERIODONTALES Y PERIIMPLANTARIAS/01/2023; TI0573) whose head is Ana María García de la Fuente, and will only be used for the purposes of this project.
Supporting Information: SAP
Time Frame: Not defined
Access Criteria: Not defined

REFERENCES:
- [Background] Landry RG, Turnbull RS, Howley T. Effectiveness of benzydamine HCl in the treatment of periodontal postsurgical patients. Research in Clinic Forums 1988;10:105-118
- [Background] Cuesta-Vargas AI, Roldan-Jimenez C, Neblett R, Gatchel RJ. Cross-cultural adaptation and validity of the Spanish central sensitization inventory. Springerplus. 2016 Oct 21;5(1):1837. doi: 10.1186/s40064-016-3515-4. eCollection 2016. PMID 27818875
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Dragovic M, Pejovic M, Stepic J, Colic S, Dozic B, Dragovic S, Lazarevic M, Nikolic N, Milasin J, Milicic B. Comparison of four different suture materials in respect to oral wound healing, microbial colonization, tissue reaction and clinical features-randomized clinical study. Clin Oral Investig. 2020 Apr;24(4):1527-1541. doi: 10.1007/s00784-019-03034-4. Epub 2019 Jul 24. PMID 31342245
- [Background] Fernandez-Jimenez A, Estefania-Fresco R, Garcia-De-La-Fuente AM, Marichalar-Mendia X, Aguirre-Zorzano LA. Description of the modified vestibular incision subperiosteal tunnel access (m-VISTA) technique in the treatment of multiple Miller class III gingival recessions: a case series. BMC Oral Health. 2021 Mar 20;21(1):142. doi: 10.1186/s12903-021-01511-5. PMID 33743644
- [Background] Ford HR, Jones P, Gaines B, Reblock K, Simpkins DL. Intraoperative handling and wound healing: controlled clinical trial comparing coated VICRYL plus antibacterial suture (coated polyglactin 910 suture with triclosan) with coated VICRYL suture (coated polyglactin 910 suture). Surg Infect (Larchmt). 2005 Fall;6(3):313-21. doi: 10.1089/sur.2005.6.313. PMID 16201941
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Tae BS, Park JH, Kim JK, Ku JH, Kwak C, Kim HH, Jeong CW. Comparison of intraoperative handling and wound healing between (NEOSORB(R) plus) and coated polyglactin 910 suture (NEOSORB(R)): a prospective, single-blind, randomized controlled trial. BMC Surg. 2018 Jul 6;18(1):45. doi: 10.1186/s12893-018-0377-4. PMID 29980202